CLINICAL TRIAL: NCT04036448
Title: Post Marketing Surveillance on Safety Evaluation of REVLIMID® (Lenalidomide) Treatment of Myelodysplastic Syndromes Associated With a Deletion 5q or Mantle Cell Lymphoma in Korea
Brief Title: A Non-interventional Study of REVLIMID® (Lenalidomide) Treatment of IPSS Low- or Intermediate-1-risk Myelodysplastic Syndromes Associated With a Deletion 5q or Refractory/Relapsed Mantle Cell Lymphoma in Korea
Acronym: RevlimidPMS
Status: Completed | Type: Observational
Sponsor: Celgene (Industry)
Responsible Party: Sponsor
Other Study IDs: CC-5013-MDS-013; U1111-1235-2858 (Other: WHO)
Record Dates: First submitted 2019-07-25; First posted 2019-07-29 (Actual); Last update posted 2025-03-11 (Actual); Status verified 2025-03

CONDITIONS: Myelodysplastic Syndromes; Lymphoma, Mantle-Cell; Lymphoma, Follicular
Keywords: REVLIMID®; Lenalidomide; Observational; Korea; Post Marketing Surveillance[PMS]; Relapsed and Refractory Mantle cell lymphoma; IPSS Low- or intermediate-1-risk Myelodysplastic Syndromes Associated with a deletion 5q; previously treated follicular lymphoma (FL) in Korea
MeSH Terms: conditions — Myelodysplastic Syndromes; Lymphoma, Mantle-Cell; Lymphoma, Follicular; Recurrence | interventions — Lenalidomide

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Lenalidomide in IPSS Low-or intermediate-1-risk del population: For the IPSS Low- or intermediate-1-risk del (5q) (MDS), Lenalidomide treatment must not be started if the ANC < 0.5 x 109/L and/or platelet counts < 25 x 109/L. The recommended starting dose of lenalidomide is 10 mg orally once daily on days 1 to 21 of repeated 28-day cycles.
  Interventions: Drug: REVLIMID®
- Lenalidomide in Refractory/relapsed rrMC/ Follicular lymphoma population: For the Refractory/relapsed Mantle cell lymphoma (rrMCL), the recommended starting dose of lenalidomide is 25 mg orally once daily on days 1 to 21 of repeated 28-day cycles. For the Follicular lymphoma (FL), the recommended starting dose of rituximab is 375 mg/m2 intravenously (IV) every week in Cycle 1 (days 1, 8, 15, and 22) and day 1 of every 28-day cycle for Cycles 2 through 5.
  Interventions: Drug: REVLIMID®

INTERVENTIONS:
Drug: REVLIMID® — REVLIMID®

SUMMARY:
The Drug Use Examination (DUE) is planned and designed for the safety evaluation of new indications after the approval of a new drug in Korea.

This DUE is a non-interventional, observational and post-marketing surveillance, which will be conducted by collecting the safety information of REVLIMID® for new indications in routine clinical practice in Korea.

Six-Hundred (600) adult patients, who start with REVLIMID® treatment based on the approved local package insert (PI) of REVLIMID® during routine clinical practice in Korea and have indications noted below.

1. Patients with transfusion-dependent anemia due to IPSS low- or intermediate-1-risk Myelodysplastic Syndromes associated with a deletion 5q cytogenetic abnormality (del [5q] MDS)
2. Patients with mantle cell lymphoma who have received at least one prior therapy (rrMCL)
3. Previously treated follicular lymphoma (FL), in combination with rituximab (an anti-CD20 antibody)

ELIGIBILITY:
Inclusion Criteria:

* Treatment of patients with transfusion-dependent anemia due to IPSS low- or intermediate-1-risk Myelodysplastic Syndromes associated with a deletion 5q cytogenetic abnormality according to International scoring system for evaluating prognosis in myelodysplastic syndromes according to IPSS or
* Treatment of patients with mantle cell lymphoma who have received at least one prior therapy
* Previously treated follicular lymphoma (FL)
* Patients who are registered in Celgene Risk Management Program" in Korea

Exclusion Criteria:

Pregnancy or females of childbearing potential

* Hypersensitivity to the active substance or to any of the excipients (e.g., angioedema, Stevens-Johnson syndrome, toxic epidermal necrolysis, DRESS)
* Patients with genetic disorder (e.g., galactose intolerance, Lapp lactase deficiency, or glucose-galactose malabsorption)

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Six-Hundred (600) adult patients, who start with REVLIMID® treatment based on the approved local package insert (PI) of REVLIMID® during routine clinical practice in Korea and have indications noted for IPSS low- or intermediate-1-risk del (5q) MDS, rrMCL and previously treated Follicular lymphoma.
Sampling Method: Non-Probability Sample
Enrollment: 28 (Actual)
Dates: Start 2019-11-28 (Actual); Primary Completion 2023-08-15 (Actual); Study Completion 2023-08-15 (Actual)

PRIMARY OUTCOMES:
Adverse events (AEs) | From enrollment until at least 28 days after completion of study treatment
  Number of participants with adverse event

SECONDARY OUTCOMES:
Adverse events (AEs) | From enrollment until at least 28 days after completion of study treatment
  Number of participants with adverse events
To evaluate the effectiveness of REVLIMID® treatment in patients with IPSS low- or intermediate-1-risk del (5q) MDS | Up to 4 years of Revlimid treatment period
  Effectiveness evaluation for IPSS low- or intermediate-1-risk del (5q) MDS is RBC transfusion-independence response rate for ≥ 56 days (8 weeks) in patients who receive at least 2 cycles of Revlimid
To evaluate the effectiveness of REVLIMID® treatment in patients with rrMCL | Up to 4 years of Revlimid treatment period
  Effectiveness evaluation for refractory/relapsed Mantle Cell Lymphoma (rrMCL) is Overall Response Rate up to 6 cycles assessed by the investigators using the Cheson Criteria, 1999
To evaluate the effectiveness of REVLIMID® treatment in patients with previously treated FL | Up to 4 years of Revlimid treatment period
  Effectiveness evaluation for refractory/relapsed previously treated FL is Overall Response Rate up to 6 cycles assessed by the investigators per 2007 International Working Group criteria.

CONTACTS AND LOCATIONS:
Overall Officials: Claire (Myoung-Jin) Lee, Medical doctor, Study Director — Celgene Korea
Locations (26):
- South Korea (26):
  - Local Institution - S02, Seoul, Seoul Teugbyeolsi
  - Hallym University Medical Center, Anyang
  - Keimyung University Dongsan Hospital, Daegu
  - Kyungpook National University Hospital, Daegu
  - Local Institution - S03, Daegu
  - Local Institution - S07, Daegu
  - Local Institution - S11, Goyang
  - CHONNAM National University Hwasun Hospital, Hwasun
  - Local Institution - S04, Hwasun-gun
  - Naitonal Health Insurance Service Ilsan hospital, Ilsan
  - Gachon University Gil Mdical Center, Incheon
  - Local Institution - S09, Incheon
  - Jeonbuk National University Hospital, Jeonju
  - Local Institution - S10, Jeonju
  - Local Institution - S05, Seoul
  - Local Institution - S06, Seoul
  - Seoul National University Hospital, Seoul
  - Local Institution - S08, Seoul
  - Yonsei University Severance Hospital, Seoul
  - Asan Medical Center, Seoul
  - Local Institution - S12, Seoul
  - Samsung Medical Center, Seoul
  - Local Institution - S01, Seoul
  - The Catholic University, St. Mary's Hospital, Seoul
  - Local Institution - S14, Wŏnju
  - Wonju Severance Christian Hospital, Wŏnju

IPD SHARING:
Plan to Share IPD: Yes
Information relating to our policy on data sharing and the process for requesting data can be found at the following link:
  https://www.celgene.com/research-development/clinical-trials/clinical-trials-data-sharing/
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: See Plan Description
Access Criteria: See Plan Description
URL: https://www.celgene.com/research-development/clinical-trials/clinical-trials-data-sharing/

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html